CLINICAL TRIAL: NCT05318638
Title: Changes in Movement Profile Related to Use of a Soft-robotic Glove During High-demand Tasks
Brief Title: Soft-robotic Glove Support of High-demand Tasks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Roessingh Research and Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 80144
Record Dates: First submitted 2021-12-21; First posted 2022-04-08 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Neuromuscular Diseases; Sarcopenia
Keywords: Soft-robotic glove; Wearable device; Hand function; Movement analysis
MeSH Terms: conditions — Neuromuscular Diseases; Sarcopenia

STUDY DESIGN:
Intervention Model Description: The study is a cross-sectional intervention study with one measurement session, where participants will perform maximum handgrip strength tests and high-demand ADL-tasks with and without the soft-robotic glove (glove condition in randomized order).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Other): All participants in the study will perform arm/hand movement tasks in both of two conditions (with and without soft-robotic glove), so they constitute 1 study arm, but all receiving both intervention conditions (experimental - with glove and control - without glove).
  Interventions: Device: Soft robotic glove

INTERVENTIONS:
Device: Soft robotic glove — The soft-robotic glove used in the study is the Carbonhand system (Bioservo Technologies, Sweden). It is a CE-marked medical device and it consists of a glove that supports finger flexion via sewn-in tendons and a control unit housing the actuators that pull on the tendons and the batteries. The grip support is activated by applying very light pressure on sensors in the fingertips of the glove, and de-activated by releasing the pressure on the sensors.

SUMMARY:
The hand is important to perform activities of daily living (ADL). However, many people experience a loss of hand function as result of a traumatic brain injury, spinal cord injury, stroke or orthopedic problems, or due to ageing. To improve hand function, or reduce its decline, one can benefit from exercise therapy or use of assistive aids to improve ADL independence. A promising innovative approach combining both is a wearable soft-robotic glove that supports hand grip. With this glove, performance of functional activities can be supported directly, while also facilitating repeated use of the affected arm and hand during functional daily activities. One of our previous studies showed that besides a direct support effect, a therapeutic effect on performance was found after several weeks of using the soft-robotic glove as support during ADL. However, several participants reported complaints of increased pain and/or overload, mainly at the beginning of the trial. Clinicians suspect that a (too) high intensity of hand use compared to normal is contributing to this observation. This might be related to more fatigue experienced when using the glove in high-demand tasks, due to a larger movement capacity (faster, further, more repetitions) and can be associated with decreased blood perfusion/lower saturation levels at muscular level and altered muscle activation and movement coordination.

Therefore, the primary objective is to examine the effect of use of the assistive soft-robotic glove during strenuous ADL tasks on the kinematic movement profile, compared to not using the soft-robotic glove. Secondary objectives are to examine whether pain or discomfort is experienced in strenuous activities with the soft-robotic glove as well as the characteristics and locations of such pain/discomfort, and to examine whether use of the glove is associated with increased handgrip strength, larger number of ADL task repetitions, diminished blood perfusion / reduced tissue saturation at the muscle and/or changes in muscle activity.

DETAILED DESCRIPTION:
A promising innovative approach to improve hand function is to integrate exercise therapy with support of activities of daily life using an assistive device. This is possible using a wearable soft-robotic glove that supports hand grip. With this glove, performance of functional activities can be supported directly, while also facilitating repeated use of the affected arm and hand during functional daily activities. One of our previous studies showed that besides a direct support effect, a therapeutic effect on performance was found after several weeks of using the soft-robotic glove as support during ADL. However, several participants reported complaints of increased pain and/or overload, mainly at the beginning of the trial. Clinicians suspect that a (too) high intensity of hand use compared to normal is contributing to this observation. This might be related to more fatigue experienced when using the glove in high-demand tasks, due to a larger movement capacity (faster, further, more repetitions) and can be associated with decreased blood perfusion/lower saturation levels at muscular level and altered muscle activation and movement coordination.

The primary objective is to examine the effect of use of the assistive soft-robotic glove during strenuous ADL tasks on the kinematic movement profile, compared to not using the soft-robotic glove. Secondary objectives are to examine whether pain or discomfort is experienced in strenuous activities with the soft-robotic glove as well as the characteristics and locations of such pain/discomfort, and to examine whether use of the glove is associated with increased handgrip strength, larger number of ADL task repetitions, diminished blood perfusion / reduced tissue saturation at the muscle and/or changes in muscle activity.

The study is set-up as a cross-sectional intervention study with one measurement session, where participants will perform maximum handgrip strength tests and high-demand ADL-tasks with and without the soft-robotic glove. The aim is to include 20 participants in total, 10 of which will be frail elderly and the other 10 will be neuromuscular patients, all suffering from reduced hand function.

All participants will perform each movement task with and without the soft-robotic glove. The soft-robotic glove used in the study is the Carbonhand system (Bioservo Technologies, Sweden). It is a CE-marked medical device and it consists of a glove that supports finger flexion via sewn-in tendons and a control unit housing the actuators that pull on the tendons and the batteries. The grip support is activated by applying very light pressure on sensors in the fingertips of the glove, and de-activated by releasing the pressure on the sensors. After execution of all tasks with and without glove, differences in outcome measures will be compared between glove conditions.

ELIGIBILITY:
Inclusion Criteria:

* Frail elderly with reduced hand function:

  * Age between 65 and 90 years
  * Experience difficulties in performing ADL due to a decline in hand function
  * Able to make a pinch grip between thumb and middle or ring finger
  * Sufficient cognitive status to understand two-step instructions
  * Having (corrected to) normal vision
  * Able to provide written informed consent
* Neuromuscular patients:

  * Age between 18 and 80 years
  * Experience difficulties in performing ADL due to a decline in hand function that can be attributed to a diagnosed neuromuscular disease
  * Being in a chronic and stable phase of disease
  * Able to make a pinch grip between thumb and middle or ring finger
  * Sufficient cognitive status to understand two-step instructions
  * Having (corrected to) normal vision
  * Able to provide written informed consent

Exclusion Criteria:

* Frail elderly with reduced hand function:

  * Currently receiving treatment for a disease affecting arm/hand function
  * Used the CarbonHand system in the past 3 months
  * Severe sensory problems of the most-affected hand
  * Severe acute pain of the most-affected hand
  * Wounds on the hands that can provide a problem when using the glove
  * Severe contractures limiting passive range of motion
  * Severe spasticity of the hand (≥2 points on Ashworth Scale)
  * Insufficient knowledge of the Dutch language to understand the purpose or methods of the study
* Neuromuscular patients:

  * Severe sensory problems of the most-affected hand

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Kinematic movement profile during performance of strenuous ADL task | 1-2 hours during the measurement session
  The kinematic movement profile during performance of strenuous ADL task, characterized by the following parameters as assessed using 3D marker-based motion capture: • Total movement duration
  * Duration of movement phases
  * Movement smoothness
  * Trunk displacement
  * Peak hand velocity
  * Time to peak velocity of reach phase
  * Hand opening
  * Joint excursion of the elbow
  * Joint excursion of the wrist
  * Endpoint straightness
  * Endpoint error

SECONDARY OUTCOMES:
Experienced pain/discomfort rating + description | Twice during the measurement session, after completion of both conditions, with a duration of 5-10 minutes.
  Discomfort and pain in the hand experienced by the participants will be assessed using a report form, indicating the amount of experienced pain and/or discomfort (using Visual Analogue Scales), and in case of discomfort or pain, a map of the hands to localize the pain/discomfort and a description of its sensation as well as an assumed cause. This will be done separately for each area in which discomfort and/or pain is reported.
Perceived exertion and confidence in grip rating | Twice during the measurement session, after completion of both conditions, with a duration of 5-10 minutes.
  Perceived exertion/fatigue after the strenuous ADL tasks will be assessed using the Borg Rating Scale of Perceived Exertion. An additional question assesses the participants' confidence in their grip on the object as experienced during the ADL task performance.
Maximal handgrip strength | 1-2 hours during the measurement session
  The maximal handgrip strength will be measured with a custom-made cylindrical dynamometer, recording the maximum force a person can exert on the dynamometer by forcefully gripping the cylinder. This will be done three times, if the last attempt is done with higher force than the second-to-last attempt, another attempt will be added, until the last value is lower than the second-to-last value.
Handgrip endurance | 1-2 hours during the measurement session
  Handgrip endurance will also be measured with a custom-made cylindrical dynamometer. It will be measured in a static situation, by prolonged max contraction of hand grip during 30 seconds.
Number of repetitions achieved during ADL task | 1-2 hours during the measurement session
  The number of repetitions achieved during execution of the ADL task (i.e., number of times the task was completed succesfully) in the four different conditions (no glove and unsupported max weight, no glove and supported max weight, glove and unsupported max weight, glove and supported max weight) will be recorded.
Muscle tissue oxygen saturation | 1-2 hours during the measurement session
  The muscle oxygen saturation in the forearm is measured during the ADL task execution and handgrip strength and endurance tests using a NIRS sensor placed over the M. flexor radialis and ulnaris and the M. flexor digitorum superficialis, secured with Velcro straps around the forearm.
Amplitude, on/off times and median frequency of muscle activity | 1-2 hours during the measurement session
  Muscle activity parameters will be calculated from surface EMG recordings of Abductor pollicis brevis, Extensor digitorum, Extensor carpi radialis, Extensor carpi ulnaris, Extensor pollicis brevis/longus, Flexor carpi ulnaris, Flexor carpi radialis

OTHER OUTCOMES:
Subject characteristics | At the start of the measurement session, taking about 5 minutes
  * Age
  * Sex
  * Most-affected side
  * Dominant side
  * Impairment/ disorder and date of diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: G. Prange, PhD, Principal Investigator — Roessingh Research and Development
Locations (1):
- Roessingh Research and Development, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No